CLINICAL TRIAL: NCT04236999
Title: Unplugged, a Drug Use Prevention Program: Adaptation and Evaluation of Effectiveness Among Students in Chile
Acronym: YSLQQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Jorge Gaete, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Fondecyt Regular 1181724
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Substance Use
Keywords: Adolescents; Unplugged; Prevention; Schools
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: In all the assessments, research assistants will be blind to the trial arm where the schools/students were allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YSLQQ group (Experimental): This group will receive the prevention program during the academic year in school hours. The prevention program is called Unplugged in its original name, but the adaptation made by the research team for Chile is called "Yo Sé Lo Que Quiero" (YSLQQ). 12 one-hour sessions taught once a week by class teachers, previously trained in a 3-day course. Each session will be delivered during the time of "Orientation" lessons.
  Interventions: Behavioral: Yo Sé Lo Que Quiero (YSLQQ)
- Control group (No Intervention): The control group will receive the usual teaching activities regarding substance use prevention.

INTERVENTIONS:
Behavioral: Yo Sé Lo Que Quiero (YSLQQ) — This program is organized in 12 sessions around three themes:
  * Knowledge and attitudes (sessions 1, 3, 5 and 9): Students reflect on their knowledge of legal and illegal drugs, using critical thinking to obtain an objective assessment of this knowledge.
  * Intrapersonal skills (sessions 4, 6, 8, 10. 11. and 12): Activities are carried out where students can put themselves in everyday situations and develop skills such as assertiveness, problem solving, among others.
  * Interpersonal skills (sessions 2 and 7): Students are instructed to practice refusal skills, assertiveness, and analyze coping strategies.
  Other Names: Unplugged
  Arms: YSLQQ group

SUMMARY:
Substance use and drug related disorders are important public health problems. Alcohol and illicit drug use account for 5.4% of the total burden of disease and the peak has been found in early adulthood (between ages 20 and 30 years). Substance use is one of the leading problems among Chilean adolescents. One out of four 8 th to 12 th graders have smoked cigarettes in the last month. A 35.6% of students (37%, girls; 34.2%, boys) between Year 8 and Year 12 have reported any alcohol use during the last month. It is worrying that a third of 14 years old students report using alcohol in the last month in Chile. Furthermore, two out of three who are using alcohol, report regularly using 5 or more drinks in a row during the last month. Cannabis use among young Chileans has increased in recent years. Today, one out of five students between Year 8 and Year 12 referred cannabis use during the last 30 days. Almost a 20% of students in Year 8 have used cannabis in the last year.

Therefore, is urgent to provide evidence-based drug preventive interventions to the Chilean population, specifically to school students, to tackle this problem and reduce the risk for a more dramatic future health scenario.

The aim of this study is to develop a culturally appropriate version of the Unplugged program to the Chilean culture, and to test its effectiveness among early adolescents in low-income primary schools in Santiago, Chile. This project involves two stages: first, formative work, where the research team will review, adapt and pilot the Spanish version of the program to Chile; and second, the culturally adapted version of Unplugged program will be tested in a single-blind two-arm cluster randomized controlled trial.

At the end of the intervention, investigators expect that students in schools receiving the Chilean version of Unplugged will have a lower proportion of substance use and a lower proportion of students passing from experimental use to regular use of tobacco, alcohol, and cannabis, than in control schools.

DETAILED DESCRIPTION:
Substance use and drug related disorders are important public health problems. Alcohol and illicit drug use account for 5.4% of the total burden of disease and the peak has been found in early adulthood (between ages 20 and 30 years). Most of substance use disorders start during adolescence, and it is well known that the earlier the use of any substance of abuse, the higher the risk for drug dependence later in life. For example, if alcohol use starts at 14 or earlier, the risk for alcohol dependence during adulthood is five or more times when compared to those individuals who start using alcohol after 21 years old.

Substance use is one of the leading problems among Chilean adolescents. One out of four 8 th to 12 th graders have smoked cigarettes in the last month. A 35.6% of students (37%, girls; 34.2%, boys) between Year 8 and Year 12 have reported any alcohol use during the last month. It is worrying that a third of 14 years old students report using alcohol in the last month in Chile. Furthermore, two out of three who are using alcohol, report regularly using 5 or more drinks in a row during the last month. Cannabis use among young Chileans has increased in recent years. Today, one out of five students between Year 8 and Year 12 referred cannabis use during the last 30 days. Almost a 20% of students in Year 8 have used cannabis in the last year.

Even though the great effort made by the Government of Chile during many years, offering several universal and targeted school-based interventions, the results are somehow frustrating. For example, the Chilean National Strategic Plan for Drugs 2003-2009 had the goal of reducing drug use in school-age population. However, during the same period cannabis and other illegal drugs use increased. Later, the Chilean National Plan for Drugs and Alcohol 2011-2014, had the goals, among school-age population, of reducing the annual prevalence of cannabis and alcohol use by 15%, and the annual prevalence of cocaine use by 10%. However, annual prevalence of cannabis use dramatically increased from 19.5% in 2011 to 34.2% in 2015; and the annual prevalence of alcohol increased from 59.3% in 2011 to 63.0% in 2015. Similar trend is seen in the annual prevalence of cocaine use, increasing from 3.2% in 2011 to 4.2% in 2015.

Therefore, is urgent to provide evidence-based drug preventive interventions to the Chilean population, specifically to school students, to tackle this problem and reduce the risk for a more dramatic future health scenario.

A recent systematic review found that the "Unplugged" program appears to have the best evidence of effectiveness, tested in several European countries. This universal school-based program targets students aged 12-14 years and aims to prevent all substance of abuse with special focus on tobacco, alcohol and marijuana. It is delivered by trained teachers in 12 sessions or units over a period of one academic year and includes teaching factual knowledge and attitudes regarding drug use (4 sessions), and training in interpersonal skills (4 sessions), and intrapersonal skills (4 sessions). No previous evaluation of this program has been carried out in Chile.

The aim of this study is to develop a culturally appropriate version of the Unplugged program to the Chilean culture, and to test its effectiveness among early adolescents in low-income primary schools in Santiago, Chile. This project involves two stages: first, formative work, where the research team will review, adapt and pilot the Spanish version of the program to Chile; and second, the culturally adapted version of Unplugged program will be tested in a single-blind two-arm cluster randomized controlled trial. This design is the most stringent design to test the effectiveness of an intervention. Investigators plan to include 37 mixed-sex schools, with a vulnerability index (School Vulnerability Index - National System of Equality Allocation (IVESINAE)) ≥ 50%, with at least two classes per Year 6 and Year 7, in each arm (Intervention vs. Control) (n=4440 students per arm). The control schools will receive the usual teaching and practice in drug prevention.

At the end of the intervention, investigators expect that students in schools receiving the Chilean version of Unplugged will have a lower proportion of substance use and a lower proportion of students passing from experimental use to regular use of tobacco, alcohol, and cannabis, than in control schools.

ELIGIBILITY:
Inclusion Criteria:

1. Schools having primary education (Year 1 to Year 8)
2. Schools located in Santiago (Chile)
3. Schools having a vulnerability index (School Vulnerability Index - National System of Equality Allocation (IVE-SINAE)) ≥ 50%*
4. Mixed-sex schools.
5. Schools having at least 2 classes in 6th and 7th grades.
6. Schools willing to participate under the conditions of the study before randomization.

   * The IVE-SINAE is built taking into account several students' and parental variables: health, family income, receiving state benefits. This percentage means the proportion of students in a school who are in most need.

Exclusion Criteria:

1. Schools having other interventions with a strong package on substance use prevention targeted the same grades.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8880 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Past month drunkenness | Past 30-day period
  Students will be asked: During the last 30 days, how many times participants have been drunk for drinking alcoholic beverages? Answers will range from "0" to "30 or more times"

SECONDARY OUTCOMES:
Weekly cigarette use | Past 7 days
  Students will be asked: How many cigarettes participants usually smoke per week? Answers will range from "0" to "20 or more cigarettes"
Past year marihuana use | Past 12-month period
  Students will be asked: How many times, during the last 12 months, participants have consumed marihuana? Answers will range from "0" to "30 or more times"
Knowledge and opinion about substance use | Past 6 months
  Students will be asked several questions regarding the Knowledge and opinion about substance use, using a validated questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Investigators plan to deposit the data collected in this study in the "UK Data Service". Data sharing will never compromise participant privacy, neither schools nor students.

REFERENCES:
- [Derived] Gaete J, Ramirez S, Gana S, Valenzuela D, Araya R. The Unplugged program in Chile ("Yo Se Lo Que Quiero") for substance use prevention among early adolescents: study protocol for a randomized controlled trial. Trials. 2022 Jan 25;23(1):76. doi: 10.1186/s13063-021-05904-3. PMID 35078522